CLINICAL TRIAL: NCT03244267
Title: Impact of a Smartphone App Reminder on Adherence Aspirin Prescribed as Anti-Thrombotic Therapy
Brief Title: App Reminder on ASA Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Association of Orthopaedic Nurses (Unknown)
Responsible Party: Principal Investigator, Deborah Wittig-Wells, RN, PhD, Adjunct Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00094970
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Thromboembolic Event
Keywords: Orthopedics
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Education (Active Comparator): Participants randomized to this arm will receive the standard education provided to patients about the importance of taking aspirin to prevent thromboembolic events after orthopedic surgery.
  Interventions: Behavioral: Standard Education
- Medication Reminder App + Standard Education (Experimental): Participants randomized to this arm will use a smartphone app with preset reminders to take aspirin to prevent thromboembolic events after orthopedic surgery in addition to usual postoperative discharge teaching.
  Interventions: Behavioral: Standard Education; Behavioral: Medication Reminder App

INTERVENTIONS:
Behavioral: Standard Education — Participants will receive the usual verbal education and printed information provided to patients about the importance of taking aspirin to prevent thromboembolic events after orthopedic surgery, medication dosage and scheduling.
Behavioral: Medication Reminder App — Participants will use a medication reminder app that is set in collaboration with the participants for times that fit into their daily lifestyle. The app will alert participants when it is time (selected by the participant) to take their medication.
  Arms: Medication Reminder App + Standard Education

SUMMARY:
The purpose of this study is to explore the impact of using a smartphone app reminder on medication adherence twice daily in adults prescribed 81 milligrams of aspirin for 35 days as anti-thrombotic therapy after knee or hip arthroplasty.

This study will randomly assign participants to get usual postoperative care which is teaching with verbal instructions and printed information about taking the aspirin at the time of discharge, or to have an app on your smartphone with preset reminders in addition to usual postoperative discharge teaching after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of using a smartphone application (app) reminder on medication adherence twice daily in 200 adults prescribed 81 milligrams of aspirin (ASA) for 35 days as anti-thrombotic therapy after knee or hip arthroplasty. The aim is to determine if an app downloaded on a smartphone that reminds patients twice a day to take their ASA as prescribed will improve ASA adherence and clinical outcomes for patients after total knee and total hip joint arthroplasty compared to those in the usual care.

This is a two group, randomized control study with random assignment into the control group for usual care or the intervention group to receive a medication reminder app for their smart phone (daily for 35 days) plus usual care. Participants will receive a baseline interview for demographic and other data and 36 day follow-up assessment, both conducted in person.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed aspirin 81 mg twice a day for 35 days
* Ability to write and speak English
* Have a smart phone with the capacity to download and set an app
* Own and use a smart phone for communication purposes

Exclusion Criteria:

* Diagnosis of mental illness
* Do not own a smart phone

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Proportion of Pills Taken | Post- Operative Visit (Day 36)
  The proportion of pills taken is defined as the percentage of pills taken by study participants.

SECONDARY OUTCOMES:
AIDS Clinical Trials Group (ACTG) Adherence Questionnaire Score | Post- Operative Visit (Day 36)
  The ACTG Adherence Questionnaire consists of 19 items measuring different aspects of efficacy (or confidence) in the management of one's medication. Each item is rated from 0 ("I cannot do at all") to 10 ("Sure I can do"), with total scores found by summing responses to individual items and dividing by 19. Higher scores correspond to higher levels of medication self-efficacy.
Aspirin (ASA) Self-Efficacy Scale Score | Post- Operative Visit (Day 36)
  The ASA Self-Efficacy Scale consists of 19 items measuring different aspects of efficacy (or confidence) in the management of one's medication. Each item is rated from 0 ("I cannot do at all") to 10 ("Sure I can do"), with total scores found by summing responses to individual items and dividing by 19. Higher scores correspond to higher levels of medication self-efficacy.
Number of Thromboembolic Events | Post- Operative Visit (Day 36)
  Clinical outcomes will be assessed at follow-up by self-report questions to ascertain if any thromboembolic events occurred.
Aspirin (ASA) General Adherence Scale Score | Post- Operative Visit (Day 36)
  The ASA General Adherence Scale measures the ease and ability to adhere to the ASA regimen as prescribed. It is scored by summing responses to the individual items and creating a total score. Higher scores indicate better self-reported adherence.
Unified Theory of Acceptance and Use of Technology (UTAUT2) Survey Score | Baseline (Pre-Intervention)
  The UTAUT2 measures antecedents (performance expectancy, effort expectancy, hedonic motivation) and behavioral intent to use mobile apps. Items are scored using a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree). Survey totals range between 14 and 112. Higher scores are indicative of greater acceptance and intent to adopt the target technology.
Performance Expectancy Subscale Score | Baseline (Pre-Intervention)
  The Performance Expectancy Subscale measures the perceived benefits of mobile app technology to the consumer. Scores range from 4 to 28, with higher totals indicating better perceptions of technology-related benefits.
Effort Expectancy Subscale Score | Baseline (Pre-Intervention)
  The Effort Expectancy Subscale measures the ease with which the consumer can learn and operate an app. Scores range from 4 to 28, with higher totals indicating greater beliefs that the technology is easy and accessible.
Hedonic Motivation Subscale Score | Baseline (Pre-Intervention)
  The Hedonic Motivation subscale measures the enjoyment, the consumer experiences from using an app. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (Absolutely True) to 7 (Absolutely Untrue). Scoring is kept continuous with higher scores indicating greater enjoyment.
Behavioral Intent Subscale Score | Baseline (Pre-Intervention)
  The Behavioral Intent Subscale measures the decision to use a mobile app. Scores range from 3 to 21, with higher totals indicating a greater intent to use or adopt an app.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Wittig-Wells, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Orthopedic and Spine Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided